CLINICAL TRIAL: NCT05554497
Title: Virtual Mindfulness-based Therapy for the Management of Endometriosis Chronic Pelvic Pain: a Novel Delivery Platform to Increase Access to Care.
Brief Title: Virtual Mindfulness for the Management of Endometriosis Pelvic Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-285C
Record Dates: First submitted 2021-04-28; First posted 2022-09-26 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Endometriosis; Chronic Pain
Keywords: Endometriosis; Chronic Pelvic Pain; Mindfulness
MeSH Terms: conditions — Endometriosis; Chronic Pain

STUDY DESIGN:
Intervention Model Description: This is a pilot project with a single arm to assess the effectiveness of a new platform to deliver a mindfulness curriculum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness training (Experimental): 8 week virtual mindfulness-based stress reduction curriculum. Weekly 2.5 hour sessions over zoom.
  Interventions: Behavioral: Mindfulness-based stress reduction curriculum

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction curriculum — Standard 8-week mindfulness-based stress reduction curriculum

SUMMARY:
Endometriosis is a gynecologic condition that can cause severe pelvic pain and significantly impair quality of life. Endometriosis symptoms cannot always be controlled by medical therapy or surgery alone, indicating a need for the development of other adjunct treatments. Mindfulness is a non-medical treatment modality that has been used in the management of chronic pelvic pain.1-3 There is preliminary data to suggest that in-person mindfulness-based workshops can also improve endometriosis-related pain, but further research is needed.4-8 There are significant barriers to utilizing in-person mindfulness resources, the largest being cost and local availability of the workshop.

The objective of this pilot project is to assess the effectiveness of virtual mindfulness-based workshops to improve quality of life and pain in patients with endometriosis. The information from the workshops will then be used to create free online resources for patients to learn mindfulness-based approaches to manage endometriosis-related pelvic pain to reduce the financial and geographical barriers to access. Better access to mindfulness-based endometriosis management will enhance the treatment options for people suffering from this condition.

DETAILED DESCRIPTION:
The objective of this pilot project is to assess the feasibility and effectiveness of virtual mindfulness-based workshops to improve quality of life and pain in patients with endometriosis. We hypothesize that virtual mindfulness-based stress reduction workshops will improve overall quality of life and decrease pain in patients with endometriosis and chronic pelvic pain. We also hypothesize that rates of narcotic pain medication use will decrease. We propose that the virtual platform will reduce some barriers to access mindfulness-based therapy.

A registered social worker with knowledge of gynecology clinic practice will create and run the virtual mindfulness workshops based on a standard mindfulness-based stress reduction curriculum. She will receive additional training in teaching mindfulness prior to the start of the study. The workshops will run weekly for eight-weeks over the Zoom platform. The sessions will last 2.5 hours and be held in the evening to ensure those with daytime commitments can participate.

For this pilot project a before and after study design will be employed. Participants will complete questionnaires before and after participation in the eight-week mindfulness workshop. Follow up questionnaires will be completed six and twelve months after completion of the workshop. The primary outcome for this study is an improvement in quality-of-life measures. Secondary outcomes are decrease in pain intensity, reduction in psychological stress, improvement in sexual function, reduction in quantity of pain modifiers used and reduction in opiate pain medication use. These main outcomes will be measured using a previously validated tool, The Endometriosis Health Profile Questionnaire (EHP-30).29 Additional tools to assess baseline demographics, barriers to accessing mindfulness and pain medication use have been created for this study. This project has been submitted to the St. Michael's Hospital research ethics board for approval.

Upon completion of the curriculum participants will be invited to a focus group to provide qualitative feedback on their experiences with mindfulness-based stress reduction, personal barriers to accessing this treatment, how it contributed to their overall treatment plan and types of activities they found mindfulness most useful for. This data will be coded by two members of the research team to look for themes and potential areas for improvements or change before proceeding with future workshops. It will also be used to inform future knowledge translation projects.

An initial 15 participants will be recruited to the study from the gynaecology clinics at St. Michael's hospital. This is a maximum group size suggested for an effective mindfulness workshop. The goal of this small group is to determine the feasibility and effectiveness of mindfulness-based therapy for endometriosis-related pelvic pain delivered in a virtual platform prior to completing a larger study.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18 and 45;
* Have been symptomatic for six months or greater;
* Clinical or surgical diagnosis of endometriosis (must have at least one of the following):

  i)Documented Clinical Diagnosis of endometriosis based on symptoms

ii)Previous endometriosis surgery confirmed by histopathology

iii)Imaging suggestive of endometriosis (ultrasound or MRI)

iv)Receiving standard medical treatment for endometriosis including combined oral contraceptives, progestin, GnRH agonists, GnRH antagonist.

Exclusion Criteria:

* Diagnosis of other chronic pain condition, other than endometriosis;
* Vulvar pain diagnosis including vulvodynia, vaginismus
* Changes to current medical treatment or surgical intervention for endometriosis during the workshop period (8 weeks) which will be reviewed at the start of each workshop session;
* Inability to attend at least 6 out of the 8-sessions;
* Inability to complete the survey package before and after the total 8-session period;
* Prior mindfulness-based workshop participation or training;
* Currently practicing mindfulness meditation.
* No internet access and microphone access: for the use of the zoom virtual platform and to enable participation in the workshops.
* Non-English speaking.
* Unable to consent.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Patients assigned female at birth are eligible to participate, current gender identity does not effect eligibility.
Enrollment: 15 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Change in Endometriosis Health Profile Questionnaire (EHP-30) | Will be done before mindfulness curriculum then upon completion of the curriculum and 6 and 12 months after curriculum.
  Validated tool to measure symptoms of endometriosis and impact on quality of life.
  Questions measured using scale: Never, Rarely, Sometimes, Often, Always. Never - never in pain or affected by it. Always - always in pain or affected by it.

SECONDARY OUTCOMES:
Change in Pain medication use | Will be done before mindfulness curriculum then upon completion of the curriculum and 6 and 12 months after curriculum.
  Questionnaire to measure pain medication use. Visual Analogue Scale.One extreme of the line represents "no pain at all" = 0, other represents "as much pain as you possibly imagine" = 10.
  Specific questions asking type of medication use - yes/no, name, frequency responses in a specified time frame (ex. in last 1 month, or 6 months).

CONTACTS AND LOCATIONS:
Locations (1):
- Unity Health Toronto - St. Michael's Hospital, Toronto, Ontario, Canada